CLINICAL TRIAL: NCT01494506
Title: A Randomized, Open Label Phase 3 Study of MM-398, With or Without 5-Fluorouracil and Leucovorin, Versus 5 Fluorouracil and Leucovorin in Patients With Metastatic Pancreatic Cancer Who Have Failed Prior Gemcitabine-based Therapy
Brief Title: Study of MM-398 With or Without 5-FU/LV, Versus 5-FU/LV in Patients With Metastatic Pancreatic Cancer
Acronym: NAPOLI-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-398-07-03-01
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic cancer; MM-398; PEP02; Metastatic pancreatic cancer; Gemcitabine refractory pancreatic cancer; Second line pancreatic cancer treatment; Pancreatic cancer post gemcitabine therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MM-398 (Experimental): MM-398 120 mg/m2 Q3W IV. Note: The published dose of ONIVYDE was expressed as the irinotecan hydrochloride trihydrate until October 2015. It is now expressed as the irinotecan free base. Converting a dose based on irinotecan hydrochloride trihydrate to a dose based on irinotecan free base is accomplished by substituting the Molecular Weight of irinotecan hydrochloride trihydrate (677.19 g/mole) with the Molecular Weight of irinotecan free base (586.68 g/mole), which results in a conversion factor of 0.866. 120 mg/m2 dose of irinotecan hydrochloride trihydrate is equivalent to 100 mg/ m2 of irinotecan free base.
  Interventions: Drug: MM-398
- 5 Fluorouracil and Leucovorin IV (Active Comparator): 5 Fluorouracil and Leucovorin IV
  Interventions: Drug: 5 Fluorouracil; Drug: Leucovorin
- MM-398, 5-FU and Leucovorin (Experimental): MM-398 80 mg/m2, 5-FU and Leucovorin Q2W IV. Note: The published dose of ONIVYDE was expressed as the irinotecan hydrochloride trihydrate until October 2015. It is now expressed as the irinotecan free base. Converting a dose based on irinotecan hydrochloride trihydrate to a dose based on irinotecan free base is accomplished by substituting the Molecular Weight of irinotecan hydrochloride trihydrate (677.19 g/mole) with the Molecular Weight of irinotecan free base (586.68 g/mole), which results in a conversion factor of 0.866. 80 mg/m2 dose of irinotecan hydrochloride trihydrate is equivalent to 70 mg/ m2 of irinotecan free base.
  Interventions: Drug: MM-398; Drug: 5 Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: MM-398 — Arm A: MM-398 120 mg/m2 IV Q3W
  Arm C: MM-398 80mg/m2 IV Q2W
  Other Names: PEP02
  Arms: MM-398; MM-398, 5-FU and Leucovorin
Drug: 5 Fluorouracil — Arm B: 5 Fluorouracil 2000 mg/m2 IV for 4 weeks followed by 2 weeks of rest every 6 weeks
  Arm C: 5 Fluorouracil 2400 mg/m2 IV every 2 weeks
  Other Names: 5-FU
  Arms: 5 Fluorouracil and Leucovorin IV; MM-398, 5-FU and Leucovorin
Drug: Leucovorin — Arm B: Leucovorin 200 mg/m2 IV for 4 weeks followed by 2 weeks of rest every 6 weeks
  Arm C: Leucovorin 400 mg/m2 IV every 2 weeks
  Other Names: Folinic Acid
  Arms: 5 Fluorouracil and Leucovorin IV; MM-398, 5-FU and Leucovorin

SUMMARY:
The study is an open label, randomized phase 3 study of MM-398 with or without 5-Fluorouracil (5-FU) and Leucovorin (also known as folinic acid), versus 5-FU and leucovorin in metastatic pancreatic cancer patients who have progressed on prior gemcitabine based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the exocrine pancreas
* Metastatic disease
* Documented disease progression after prior gemcitabine based therapy
* KPS >/= 70
* Adequate bone marrow function
* Adequate hepatic function
* Adequate renal function

Exclusion Criteria:

* Active CNS metastasis
* Clinically significant GI disorders
* Severe arterial thromboembolic events less than 6 months before inclusion
* NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure
* Active infection or uncontrolled fever
* Pregnant or breast feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eliel Bayever, MD, Study Director — Merrimack Pharmaceuticals
Locations (79):
- United States (23):
  - Gilbert, Arizona
  - Glendale, Arizona
  - Scottsdale, Arizona
  - Burbank, California
  - Duarte, California
  - Fresno, California
  - LaVerne, California
  - San Luis Obispo, California
  - Boyton Beach, Florida
  - Atlanta, Georgia
  - Kansas City, Missouri
  - St Louis, Missouri
  - Henderson, Nevada
  - Albuquerque, New Mexico
  - Buffalo, New York
  - Columbus, Ohio
  - Norman, Oklahoma
  - Greenville, South Carolina
  - Bedford, Texas
  - Dallas, Texas
  - Tyler, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
- Argentina (3):
  - Buenos Aires
  - Rosario
  - Santa Fe
- Australia (6):
  - Westmead, New South Wales
  - Kurralta Park, South Australia
  - Boxhill, Victoria
  - Heidelberg, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
- Brazil (5):
  - Belo Horizonte
  - Ijuí
  - Passo Fundo
  - Porto Alegre
  - São Paulo
- Montreal, Quebec, Canada
- Czechia (4):
  - Hořovice
  - Olomouc
  - Prague
  - Příbram
- France (3):
  - Bordeaux
  - Lille
  - Marseille
- Germany (4):
  - Berlin
  - Jens
  - Munich
  - Ulm
- Hungary (5):
  - Budapest
  - Pécs
  - Szeged
  - Szolnok
  - Szombathely
- Italy (5):
  - Castellana Grotte
  - Genova
  - Legnano
  - Naples
  - Roma
- South Africa (3):
  - Port Elizabeth
  - Pretoria
  - Western Cape
- South Korea (2):
  - Hwasun-gun
  - Seoul
- Spain (5):
  - Alicante
  - Barcelona
  - Madrid
  - Santander
  - Valencia
- Taiwan (6):
  - Chiayi City
  - Kaohsiung City
  - Taiching
  - Tainan
  - Taipei
  - Taoyuan District
- United Kingdom (4):
  - Liverpool
  - London
  - Manchester
  - Sutton

REFERENCES:
- [Derived] Chen LT, Macarulla T, Blanc JF, Mirakhur B, de Jong FA, Belanger B, Bekaii-Saab T, Siveke JT. Early dose reduction/delay and the efficacy of liposomal irinotecan with fluorouracil and leucovorin in metastatic pancreatic ductal adenocarcinoma (mPDAC): A post hoc analysis of NAPOLI-1. Pancreatology. 2021 Jan;21(1):192-199. doi: 10.1016/j.pan.2020.10.029. Epub 2020 Oct 10. PMID 33214082
- [Derived] Macarulla Mercade T, Chen LT, Li CP, Siveke JT, Cunningham D, Bodoky G, Blanc JF, Lee KH, Dean A, Belanger B, Wang-Gillam A. Liposomal Irinotecan + 5-FU/LV in Metastatic Pancreatic Cancer: Subgroup Analyses of Patient, Tumor, and Previous Treatment Characteristics in the Pivotal NAPOLI-1 Trial. Pancreas. 2020 Jan;49(1):62-75. doi: 10.1097/MPA.0000000000001455. PMID 31856081
- [Derived] Bang YJ, Li CP, Lee KH, Chiu CF, Park JO, Shan YS, Kim JS, Chen JS, Shim HJ, Rau KM, Choi HJ, Oh DY, Belanger B, Chen LT. Liposomal irinotecan in metastatic pancreatic adenocarcinoma in Asian patients: Subgroup analysis of the NAPOLI-1 study. Cancer Sci. 2020 Feb;111(2):513-527. doi: 10.1111/cas.14264. Epub 2019 Dec 20. PMID 31789476
- [Derived] Macarulla T, Blanc JF, Wang-Gillam A, Chen LT, Siveke JT, Mirakhur B, Chen J, de Jong FA. Liposomal irinotecan and 5-fluorouracil/leucovorin in older patients with metastatic pancreatic cancer - A subgroup analysis of the pivotal NAPOLI-1 trial. J Geriatr Oncol. 2019 May;10(3):427-435. doi: 10.1016/j.jgo.2019.02.011. Epub 2019 Mar 4. PMID 30842038
- [Derived] Wang-Gillam A, Hubner RA, Siveke JT, Von Hoff DD, Belanger B, de Jong FA, Mirakhur B, Chen LT. NAPOLI-1 phase 3 study of liposomal irinotecan in metastatic pancreatic cancer: Final overall survival analysis and characteristics of long-term survivors. Eur J Cancer. 2019 Feb;108:78-87. doi: 10.1016/j.ejca.2018.12.007. Epub 2019 Jan 14. PMID 30654298
- [Derived] Chen LT, Siveke JT, Wang-Gillam A, Li CP, Bodoky G, Dean AP, Shan YS, Jameson GS, Macarulla T, Lee KH, Cunningham D, Blanc JF, Chiu CF, Schwartsmann G, Braiteh FS, Mamlouk K, Belanger B, de Jong FA, Hubner RA. Survival with nal-IRI (liposomal irinotecan) plus 5-fluorouracil and leucovorin versus 5-fluorouracil and leucovorin in per-protocol and non-per-protocol populations of NAPOLI-1: Expanded analysis of a global phase 3 trial. Eur J Cancer. 2018 Dec;105:71-78. doi: 10.1016/j.ejca.2018.09.010. Epub 2018 Nov 8. PMID 30414528
- [Derived] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized over a period of 1.9 years starting from 2012-01-11 to 2013-09-11.
  The study was initially a two-arm study with MM-398 monotherapy and 5-FU/LV control (protocol version 1) . A third arm of MM-398+5-FU/LV was added later (protocol version 2).
Pre-assignment Details: All patients were screened for UGT1A1*28 allele at baseline.
Groups:
- MM-398 (Arm A): • MM-398 120 mg/m2 IV on Day 1of a 3 weekly cycle Patients who were homozygous for UGT1A1*28 allele received the first cycle of therapy at a reduced dose of 80 mg/m2. If the patient did not experience any drug related toxicity after the first administration of MM-398, from cycle 2 onwards, the dose could be increased in increments of 20 mg/m2 up to a maximum of 120 mg/m2.
- 5-FU + Leucovorin (Arm B): * 5-FU 2000 mg/m2 IV over 24-hours, every week for 4 weeks (days 1, 8, 15 and 22), followed by 2 weeks of rest, in a 6 week cycle
  * Leucovorin l + d racemic form 200 mg/m2, or l form 100 mg/m2 IV over 30 minutes, every week for 4 weeks (days 1, 8, 15 and 22), followed by 2 weeks of rest, in a 6 week cycle.
- MM-398 + 5-FU + Leucovorin (Arm C): * MM-398 80 mg/m2 IV every 2 weeks Patients who were homozygous for UGT1A1*28 allele and were randomized to Arm C, received the first cycle of therapy at a reduced dose of 60 mg/m2. If the patient did not experience any drug related toxicity after the first administration of MM-398, from cycle 2 onwards, the dose could be increased to 80 mg/m2.
  * 5-FU 2400 mg/m2 IV over 46-hours, and
  * Leucovorin l + d racemic form 400 mg/m2, or l form 200 mg/m2 IV over 30 minutes, every 2 weeks
Period: Overall Study
Arm/Group | MM-398 (Arm A) | 5-FU + Leucovorin (Arm B) | MM-398 + 5-FU + Leucovorin (Arm C)
Started | 151 (Started = Intent to Treat Population and includes all randomized participants) | 149 | 117
Treated Population | 147 (Treated population: Patients who received at least 1 dose of study drug.) | 134 | 117 (2 randomized Arm C patients did not receive study drug. 1 patient each in A and B received Arm C.)
Completed | 3 (Completed = Subjects remaining on treatment at the time of the primary analysis data cut off.) | 6 | 14
Not Completed | 148 | 143 | 103
Not completed — Lack of Efficacy | 77 | 83 | 57
Not completed — Adverse Event | 17 | 10 | 11
Not completed — Death | 9 | 5 | 2
Not completed — Physician Decision | 7 | 5 | 4
Not completed — Withdrawal by Subject | 17 | 20 | 14
Not completed — Clinical Deterioration | 21 | 17 | 13
Not completed — Sponsor Decision | 0 | 0 | 1
Not completed — Other | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients.
Groups:
- MM-398: MM-398 Q3W IV
  MM-398: Arm A: MM-398 120 mg/m2 IV Q3W
  Arm C: MM-398 80mg/m2 IV Q2W
- 5 Fluorouracil and Leucovorin IV: 5 Fluorouracil and Leucovorin IV
  5 Fluorouracil: Arm B: 5 Fluorouracil 2000 mg/m2 IV for 4 weeks followed by 2 weeks of rest every 6 weeks
  Arm C: 5 Fluorouracil 2400 mg/m2 IV every 2 weeks
  Leucovorin: Arm B: Leucovorin 200 mg/m2 IV for 4 weeks followed by 2 weeks of rest every 6 weeks
  Arm C: Leucovorin 400 mg/m2 IV every 2 weeks
- MM-398, 5-FU and Leucovorin: MM-398, 5-FU and Leucovorin Q2W IV
  MM-398: Arm A: MM-398 120 mg/m2 IV Q3W
  Arm C: MM-398 80mg/m2 IV Q2W
  5 Fluorouracil: Arm B: 5 Fluorouracil 2000 mg/m2 IV for 4 weeks followed by 2 weeks of rest every 6 weeks
  Arm C: 5 Fluorouracil 2400 mg/m2 IV every 2 weeks
  Leucovorin: Arm B: Leucovorin 200 mg/m2 IV for 4 weeks followed by 2 weeks of rest every 6 weeks
  Arm C: Leucovorin 400 mg/m2 IV every 2 weeks
- Total: Total of all reporting groups
Arm/Group | MM-398 | 5 Fluorouracil and Leucovorin IV | MM-398, 5-FU and Leucovorin | Total
Number analyzed (Participants) | 151 | 149 | 117 | 417
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 151 | 149 | 117 | 417
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (10.13) | 61.8 (9.65) | 63.2 (9.06) | 62.8 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 48 | 180
  Male | 87 | 81 | 69 | 237
RACE (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 52 | 50 | 34 | 136
  Black or African American | 3 | 3 | 4 | 10
  White | 89 | 92 | 72 | 253
  other race | 6 | 4 | 7 | 17
Karnofsky Performance Status (Baseline KPS)[1] [Number; unit: participants] — 1. One patient in the 5-FU/LV arm did not have a recorded Baseline KPS value.
  2. Designation of the KPS level for the randomization strata is made during the screening period prior to knowledge of the treatment assignment. Baseline KPS is the last observed KPS value prior to treatment in treated patients and the last observed value in patients who were randomized and did not receive study drug. The observed baseline KPS value may be recorded post-randomization.
  participants
    100% = normal, no complaints, no signs of disease | 22 | 22 | 18 | 62
    90% = normal activity, few symptoms of disease | 64 | 54 | 51 | 169
    80% = normal activity, some symptoms of disease | 50 | 61 | 38 | 149
    70% = caring for self, unable to work | 15 | 11 | 7 | 33
    60% [2] = needs help, can manage most tasks | 0 | 0 | 2 | 2
    50%[2]= needs help often and medical care | 0 | 0 | 1 | 1
    Not recorded | 0 | 1 | 0 | 1
Pancreatic Primary Tumor Location [Number; unit: participants]
  Head | 92 | 77 | 70 | 239
  Body | 16 | 26 | 12 | 54
  Tail | 24 | 24 | 14 | 62
  Multiple locations including head | 7 | 4 | 6 | 17
  Multiple locations not including head | 7 | 14 | 9 | 30
  Unknown = not specified | 5 | 4 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was the primary efficacy endpoint of the study and was defined as the time from the date of patient randomization to the date of death or the date the patient was last known to be alive. OS was summarized by Kaplan-Meier methodology for each treatment group. Pairwise treatment group comparisons were carried out using unstratified log rank analyses on the ITT population. Hazard ratio estimates are from Cox regression analysis.
  The comparison of Arm C is based only on patients who were randomized under the 3-arm version of the protocol. Consequently, the 5-FU+Leucovorin (Combo Therapy Comparison) group is a subset of all patients randomized to 5-FU+Leucovorin, which is the Mono Therapy Comparison control and contains patients randomized under both the 2-arm and 3-arm versions of the protocol.
Time Frame: From randomization to death; until the data cut off 14 Feb 2014. The maximum time in follow up was 25 months.
Population: Intent to Treat population (ITT population) consisted of all randomized participants. Efficacy analyses in the ITT population consider treatment group according to randomization. Comparisons of the MM-398+5-FU/LV to 5-FU/LV were carried out only on patients who were randomized under protocol version 2 or later.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- MM-398 Arm A (Mono Therapy Comparison): • MM-398 120 mg/m2 IV on Day 1of a 3 weekly cycle Patients who were homozygous for UGT1A1*28 allele received the first cycle of therapy at a reduced dose of 80 mg/m2. If the patient did not experience any drug related toxicity after the first administration of MM-398, from cycle 2 onwards, the dose could be increased in increments of 20 mg/m2 up to a maximum of 120 mg/m2.
- 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); 5-FU + Leucovorin (Combo Therapy Comparison): * 5-FU 2000 mg/m2 IV over 24-hours, every week for 4 weeks (days 1, 8, 15 and 22), followed by 2 weeks of rest, in a 6 week cycle
  * Leucovorin l + d racemic form 200 mg/m2, or l form 100 mg/m2 IV over 30 minutes, every week for 4 weeks (days 1, 8, 15 and 22), followed by 2 weeks of rest, in a 6 week cycle.
- MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison: * MM-398 80 mg/m2 IV every 2 weeks Patients who were homozygous for UGT1A1*28 allele and were randomized to Arm C, received the first cycle of therapy at a reduced dose of 60 mg/m2. If the patient did not experience any drug related toxicity after the first administration of MM-398, from cycle 2 onwards, the dose could be increased to 80 mg/m2.
  * 5-FU 2400 mg/m2 IV over 46-hours, and
  * Leucovorin l + d racemic form 400 mg/m2, or l form 200 mg/m2 IV over 30 minutes, every 2 weeks
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 151 | 149 | 117 | 119
months | 4.9 [4.23 to 5.62] | 4.2 [3.58 to 4.86] | 6.1 [4.76 to 8.87] | 4.2 [3.29 to 5.32]
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Test type: Superiority or Other; p = 0.9416, Log Rank; Unstratified logrank test; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.77 to 1.28]
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Test type: Superiority or Other; p = 0.012, Log Rank; Unstratified logrank test; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.49 to 0.92]

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival was defined as the time from the date of randomization to the date of disease progression, or death (any cause) on or prior to the clinical cutoff date, whichever occurred earlier. Participants who did not have disease progression or had not died were censored at the date of the last tumor assessment. Patients with two or more consecutive missing response assessments prior to a visit with documented progression (or death) were censored at the last date of tumor assessment when the patient was documented to be progression free. PFS was summarized using Kaplan-Meier methods.
  The comparison of Arm C is based only on patients who were randomized under the 3-arm version of the protocol. Consequently, the 5-FU+Leucovorin (Combo Therapy Comparison) group is a subset of all patients randomized to 5-FU+Leucovorin, which is the Mono Therapy Comparison control and contains patients randomized under both the 2-arm and 3-arm versions of the protocol.
Time Frame: Randomization until disease progression or death from any cause; Until the data cut off of 14 Feb 2014. The maximum time in follow up was 25 months.
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 151 | 149 | 117 | 119
months | 2.7 [2.13 to 2.89] | 1.6 [1.41 to 1.84] | 3.1 [2.69 to 4.17] | 1.5 [1.41 to 1.84]
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Test type: Superiority or Other; p = 0.100, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.63 to 1.04]
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Test type: Superiority or Other; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.41 to 0.75]

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate was a secondary efficacy endpoint of the study and was defined by the percentage of patients in the study population with a best overall response of Complete Response (CR) or Partial Response (PR) as assessed by the investigator. Best overall response was defined per RECIST (version 1.1) recorded from randomization until progression or end of study. RECIST (v 1.1) criteria does not require confirmation of response, but an additional, more stringent analysis was also conducted, with designation of CR (or PR) requiring confirmation of response at least 4 weeks following the initial assessment of CR (or PR). Stable disease (SD) required an assessment of SD at least 6 weeks after starting treatment. Subjects with insufficient data for response classification were classified as Not Evaluable for best overall response, and as a non-responder for objective response, in the ITT population. Treatment groups are as indicated for the primary outcome of OS.
Time Frame: Assessment every 6 weeks after initial response; Day 1 to data cut off of 14 Feb 2014; maximum time on study 25 months.
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage with confirmed response
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 151 | 149 | 117 | 119
percentage with confirmed response | 3.31 [0.46 to 6.17] | 0.67 [0.0 to 1.98] | 7.69 [2.86 to 12.52] | 0.84 [0.0 to 2.48]
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Test type: Superiority or Other; p = 0.214, Fisher Exact; Risk Difference (RD) = 0.0264, 95% CI 2-sided [-0.005 to 0.058]
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Test type: Superiority or Other; p = 0.010, Fisher Exact; Risk Difference (RD) = 0.069, 95% CI 2-sided [0.018 to 0.120]

4. Secondary Outcome: Time to Treatment Failure
Description: Time from randomization to discontinuation of treatment for any reason, including disease progression, treatment toxicity or death.
Time Frame: Randomization to treatment discontinuation (any cause). The maximum time in follow up was 25 months
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 151 | 149 | 117 | 119
months | 1.7 [1.5 to 2.7] | 1.4 [1.3 to 1.4] | 2.3 [1.6 to 2.8] | 1.4 [1.3 to 1.4]
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Test type: Superiority or Other; p = 0.1008, Log Rank; Unstratified log rank test; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.03]
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Test type: Superiority or Other; p = 0.0002, Log Rank; Unstratified log rank test; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.45 to 0.78]

5. Secondary Outcome: Percentage of Patients With Clinical Benefit Response
Description: Composite measure based on patient-reported pain (per VAS), patient-reported pain medication, KPS, and weight. Clinical benefit is indicated by either:
  (a) improvement in pain (less pain intensity with stable or decreased pain medication; or less pain medication with stable or decreased pain intensity) with stable or improved KPS; or (b) improvement in KPS with stable or improved pain.
  With stable for KPS and pain, clinical benefit may be indicated with an observation of positive weight change.
  Clinical benefit response (CBR) was classified weekly and a patient was considered a clinical benefit responder if clinical benefit was observed and maintained over a 4 week period.
Time Frame: Randomization to treatment discontinuation.The maximum time in follow up was 25 months
Population: Clinical Benefit Response Evaluable Population: Patients who received study drug and met at least one of the following criteria were defined as eligible for evaluation of CBR:
  * baseline pain intensity ≥ 20 (out of 100)
  * baseline morphine consumption ≥ 10 mg/day PO morphine equivalents
  * baseline KPS of 70 to 90 points
Measure: Number; unit: percentage of participants with CBR
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 92 | 80 | 78 | 60
percentage of participants with CBR | 14 | 13 | 14 | 12
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Test type: Superiority or Other; p = 0.82, Fisher Exact
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Test type: Superiority or Other; p = 0.80, Fisher Exact

6. Secondary Outcome: Percentage of Patients With Tumor Marker (CA 19-9) Response
Description: Tumor marker response (TMR) was evaluated by the change in CA19-9 serum levels. Response was defined as a decrease of 50% of CA19-9 in relation to the baseline level at least once during the treatment period.
Time Frame: Baseline to treatment discontinuation every 6 weeks; The maximum time in follow up was 25 months
Population: Patients with elevated baseline CA19-9 value (> 30 U/mL) who received study drug.
Measure: Number; unit: percent of participants with TMR
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 123 | 105 | 97 | 81
percent of participants with TMR | 23.6 | 11.4 | 28.9 | 8.6
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Test type: Superiority or Other; p = 0.024, Fisher Exact
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Test type: Superiority or Other; p < 0.001, Fisher Exact

7. Secondary Outcome: EORTC-QLQ-C30
Description: This patient recorded outcome consists of 15 subscales in 3 independent domains: global health-related quality of life (HRQoL), functional scales (cognitive, emotional, physical, role and social functioning), and symptom scales (appetite loss, constipation, diarrhea, dyspnea, fatigue, insomnia, nausea and vomiting, and pain). For each subscale, patients were classified as improved, worsened or stable. Improvement is indicated by achievement of subscale score at least 10% improved from baseline and maintained for at least 6 weeks. Worsened is indicated by subscale score at least 10% worse than baseline. Stable is indicated by neither improvement nor worsened. Achievement of improvement prior to worsening was classified as improvement.
Time Frame: Baseline to treatment discontinuation every 6 weeks; The maximum time in follow up was 25 months
Population: ITT patients who had baseline and at least one-post baseline EORTC-QLQ-C30 assessment.
Measure: Number; unit: percent of patients in category
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison | 5-FU + Leucovorin (Combo Therapy Comparison)
Number analyzed (Participants) | 105 | 83 | 71 | 57
percent of patients in category
  Global Health Status: Improved | 10 | 11 | 17 | 12
  Global Health Status: Stable | 31 | 41 | 38 | 44
  Global Health Status: Worsened | 57 | 48 | 45 | 44
  Physical Functioning: Improved | 10 | 11 | 10 | 11
  Physical Functioning: Stable | 29 | 37 | 41 | 40
  Physical Functioning: Worsened | 61 | 52 | 49 | 49
  Role Functioning: Improved | 6 | 10 | 15 | 11
  Role Functioning: Stable | 29 | 39 | 32 | 37
  Role Functioning: Worsened | 66 | 52 | 52 | 53
  Emotional Functioning:Improved | 10 | 8 | 20 | 9
  Emotional Functioning:Stable | 32 | 59 | 46 | 58
  Emotional Functioning:Worsened | 56 | 33 | 34 | 33
  Cognitive Functioning:Improved | 12 | 6 | 11 | 7
  Cognitive Functioning:Stable | 32 | 42 | 48 | 44
  Cognitive Functioning:Worsened | 54 | 52 | 41 | 49
  Social Functioning:Improved | 11 | 11 | 13 | 11
  Social Functioning:Stable | 26 | 43 | 34 | 47
  Social Functioning:Worsened | 62 | 46 | 54 | 42
  Fatigue:Improved | 13 | 11 | 14 | 12
  Fatigue:Stable | 18 | 30 | 20 | 33
  Fatigue:Worsened | 69 | 59 | 66 | 54
  Nausea and Vomiting:Improved | 5 | 6 | 13 | 4
  Nausea and Vomiting:Stable | 37 | 42 | 32 | 46
  Nausea and Vomiting:Worsened | 58 | 52 | 55 | 51
  Pain:Improved | 20 | 10 | 27 | 11
  Pain:Stable | 30 | 37 | 34 | 40
  Pain:Worsened | 50 | 53 | 39 | 49
  Dyspnoea:Improved | 10 | 6 | 7 | 5
  Dyspnoea:Stable | 47 | 69 | 51 | 68
  Dyspnoea:Worsoned | 44 | 24 | 42 | 25
  Insomnia:Improved | 9 | 4 | 18 | 5
  Insomnia:Stable | 43 | 49 | 34 | 49
  Insomnia:Worsened | 48 | 47 | 48 | 46
  Appetite Loss:Improved | 9 | 6 | 11 | 5
  Appetite Loss:Stable | 38 | 42 | 45 | 46
  Appetite Loss:Worsened | 53 | 52 | 44 | 49
  Constipation:Improved | 13 | 4 | 13 | 4
  Constipation:Stable | 47 | 63 | 56 | 67
  Constipation:Worsened | 39 | 34 | 31 | 30
  Diarrhoea:Improved | 4 | 4 | 6 | 4
  Diarrhoea: Stable | 35 | 58 | 39 | 58
  Diarrhoea: Worsened | 59 | 39 | 55 | 39
  Financial Difficulties: Improved | 6 | 1 | 8 | 0
  Financial Difficulties: Stable | 51 | 67 | 51 | 74
  Financial Difficulties: Worsened | 42 | 31 | 41 | 26
Statistical Analysis 1: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Global Health Status; Test type: Superiority or Other; p = 0.6388, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 2: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison; Comparison of Global Health Status; Test type: Superiority or Other; p = 0.8445, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 3: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Physical Functioning; Test type: Superiority or Other; p = 0.6388, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 4: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Physical Functioning; Test type: Superiority or Other; p = 0.9435, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 5: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Role functioning; Test type: Superiority or Other; p = 0.2654, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 6: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Role functioning; Test type: Superiority or Other; p = 0.7674, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 7: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Emotional Functioning; Test type: Superiority or Other; p = 0.1628, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 8: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Emotional Functioning; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 9: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Cognitive Functioning; Test type: Superiority or Other; p = 0.7738, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 10: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Cognitive Functioning; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 11: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Social Functioning; Test type: Superiority or Other; p = 0.3408, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 12: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Social Functioning; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 13: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Fatigue; Test type: Superiority or Other; p = 0.6766, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 14: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Fatigue; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 15: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Nausea and Vomiting; Test type: Superiority or Other; p = 0.6388, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 16: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Nausea and Vomiting; Test type: Superiority or Other; p = 0.7674, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 17: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Pain; Test type: Superiority or Other; p = 0.4993, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 18: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Pain; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 19: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Dyspnoea; Test type: Superiority or Other; p = 0.2654, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 20: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Dyspnoea; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 21: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Insomnia; Test type: Superiority or Other; p = 0.7617, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 22: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Insomnia; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel
Statistical Analysis 23: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Appetite loss; Test type: Superiority or Other; p = 0.9123, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 24: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Appetite loss; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 25: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Constipation; Test type: Superiority or Other; p = 0.7617, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 26: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Constipation; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 27: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Diarrhoea; Test type: Superiority or Other; p = 0.1628, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 28: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Diarrhoea; Test type: Superiority or Other; p = 0.6712, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 29: Comparison: MM-398 Arm A (Mono Therapy Comparison) vs 5-FU + Leucovorin (Arm B) (Mono Therapy Comparison); Comparison of Financial difficulties; Test type: Superiority or Other; p = 0.6388, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method
Statistical Analysis 30: Comparison: MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison vs 5-FU + Leucovorin (Combo Therapy Comparison); Comparison of Financial difficulties; Test type: Superiority or Other; p = 0.7308, Cochran-Mantel-Haenszel — For each experimental arm comparison p-values were adjusted for multiple domain comparisons using the Hochberg method

8. Secondary Outcome: Pharmacokinetic Measurements of Total Irinotecan
Description: Plasma concentration-time data for MM-398 will be analyzed using population pharmacokinetic methods.
Time Frame: 6 weeks after first study drug administration
Population: PK population was based on Protocol, all participants who received the appropriate dose of MM-398.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Total irinotecan = ug/L; SN38= ug/L
Arm/Group | MM-398 Arm A (Mono Therapy Comparison) | MM-398 + 5-FU + Leucovorin(Arm C) Combo Therapy Comparison
Number analyzed (Participants) | 143 | 114
Total irinotecan = ug/L; SN38= ug/L
  Total Irinotecan-Cavg | 2550.00 (197.4) | 2120.00 (209.7)
  Total Irinotecan-Cmax | 40550.00 (172.3) | 28460.00 (69.3)
  Total SN38-Cavg | 0.82 (119.2) | 0.68 (132.7)
  Total SN38-Cmax | 3.93 (119.6) | 2.58 (121.9)

ADVERSE EVENTS:
Time Frame: Study drug initiation through 30 days after the last dose of study drug or EOS, whichever is later; Up to 764 days.
Description: 5-FU= 5-fluorouracil; LV=leucovorin Events were collected by systematic assessment Term from vocabulary, MedDRA version 14.1
Arm/Group | MM-398 | 5 Fluorouracil and Leucovorin IV | MM-398, 5-FU and Leucovorin
Serious Adverse Events (participants affected / at risk) | 90/147 | 58/134 | 56/117
Other Adverse Events (participants affected / at risk) | 145/147 | 132/134 | 116/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MM-398 (N=147) | 5 Fluorouracil and Leucovorin IV (N=134) | MM-398, 5-FU and Leucovorin (N=117)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 6 | 6 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 19 | 2 | 7
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 2
Gastro Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 4
Small Intestinal Obstruction (Gastrointestinal disorders) | 3 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 14 | 2 | 11
Asthenia (General disorders) | 2 | 1 | 2
General Physical Health Deterioration (General disorders) | 3 | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 5 | 2 | 3
Bile Duct Obstruction (Hepatobiliary disorders) | 2 | 2 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 2 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 2 | 0 | 0
Biliary Tract Infection (Infections and infestations) | 1 | 2 | 2
Clostridium Difficile Colitis (Infections and infestations) | 2 | 0 | 0
Device Related Infection (Infections and infestations) | 1 | 0 | 3
Gastroenteritis (Infections and infestations) | 2 | 0 | 2
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 3
Sepsis (Infections and infestations) | 3 | 1 | 4
Septic Shock (Infections and infestations) | 3 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2 | 1
Decrease Appetite (Metabolism and nutrition disorders) | 6 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 3
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 2 | 1
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 0 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 2 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 2 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MM-398 (N=147) | 5 Fluorouracil and Leucovorin IV (N=134) | MM-398, 5-FU and Leucovorin (N=117)
Diarrhoea (Gastrointestinal disorders) | 103 | 35 | 116
Vomiting (Gastrointestinal disorders) | 80 | 35 | 61
Nausea (Gastrointestinal disorders) | 89 | 46 | 60
Decreased Appetite (Metabolism and nutrition disorders) | 72 | 43 | 52
Fatigue (General disorders) | 54 | 37 | 47
Anaemia (Blood and lymphatic system disorders) | 48 | 31 | 44
Abdominal Pain (Gastrointestinal disorders) | 50 | 42 | 27
Pyrexia (General disorders) | 29 | 15 | 27
Neutropenia (Blood and lymphatic system disorders) | 22 | 4 | 27
Constipation (Gastrointestinal disorders) | 26 | 32 | 26
Asthenia (Gastrointestinal disorders) | 35 | 22 | 24
Weight Decreased (General disorders) | 29 | 9 | 20
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 15 | 2 | 17
White Blood Cell Count Decreased (Blood and lymphatic system disorders) | 10 | 2 | 17
Alopecia (General disorders) | 32 | 6 | 16
Stomatitis (Gastrointestinal disorders) | 5 | 8 | 16
Dizziness (General disorders) | 17 | 13 | 15
Back Pain (General disorders) | 12 | 16 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 12 | 14
Oedema Peripheral (General disorders) | 28 | 20 | 13
Mucosal Inflammation (Hepatobiliary disorders) | 8 | 5 | 12
Leukopenia (Blood and lymphatic system disorders) | 6 | 1 | 12
Platelet Count Decreased (Blood and lymphatic system disorders) | 3 | 3 | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 17 | 10 | 11
Abdominal Distension (Gastrointestinal disorders) | 12 | 8 | 10
Dehydration (Metabolism and nutrition disorders) | 15 | 9 | 9
Insomnia (General disorders) | 12 | 5 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 9
Mouth Ulceration (General disorders) | 6 | 3 | 8
Alanine Aminotransferase Increased (Investigations) | 5 | 2 | 8
Hypomagnesaemia (Investigations) | 20 | 5 | 7
Hypoalbumineamia (Metabolism and nutrition disorders) | 19 | 8 | 7
Hypotension (General disorders) | 6 | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 6
Headache (General disorders) | 8 | 6 | 6
Oral Candidiasis (Infections and infestations) | 4 | 2 | 6
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 6 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 9 | 5
Ascites (Gastrointestinal disorders) | 14 | 11 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 3 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 4 | 3
Aspartate Aminotransferase Increased (Investigations) | 9 | 3 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 8 | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship/contents of any publication is determined by site and provides sponsor a publication prior to submission. Sponsor has 60 days to review and avoid editorial changes but may request site delete confidential data. If publication contains patentable matter, site agrees to delay publication for 60 days. If study is part of multicenter protocol, site agrees not to independently publish. If multicenter publication is not forthcoming in 18 months after study end, site may proceed accordingly.